CLINICAL TRIAL: NCT00615537
Title: Pilot Study on Laser Ablation of Symptomatic Benign Thyroid Masses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BioTex, Inc. (Industry)
Collaborators: Rhode Island Hospital (Other)
Responsible Party: Ashok Gowda, Ph.D. President, BioTex, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTX-07-003
Record Dates: First submitted 2008-02-03; First posted 2008-02-14 (Estimated); Last update posted 2011-04-05 (Estimated); Status verified 2011-04

CONDITIONS: Thyroid Nodule; Thyroid Cancer; Thyroid Neoplasms; Nodular Goiter
Keywords: Thyroid Nodule; Thyroid Cancer; Laser Ablation; LITT; Nodular Goiter; Thyroid Mass
MeSH Terms: conditions — Thyroid Nodule; Thyroid Neoplasms; Goiter, Nodular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Laser Ablation of Thyroid Nodule — Laser ablation using a laser generator, disposable fiberoptic laser fiber, cooling catheter and pump, will be performed under conscious sedation. Ultrasound will be used to localize masses. Local anesthesia will be administered both intradermally and subcutaneously. The laser applicator will be placed into the mass and laser energy will be delivered at 15W for 30-120 seconds. Real-time ultrasound monitoring of the ablation front will be used to ensure complete treatment of the target lesion. In larger masses applicators may be placed of the applicator into multiple locations. The number of locations will be determined by the treatment team, and based on lesion morphology, size, location, and accessibility.
  Other Names: PhoTex15 Diode Laser; Visualase Cooled Laser Applictor System

SUMMARY:
This proposal is designed as a pilot study for the use of laser ablation for local control of symptomatic (e.g compressive) benign thyroid masses in 20 patients.

DETAILED DESCRIPTION:
Thyroid nodules are a very common clinical finding, with an estimated prevalence (based on palpation) ranging from 3% to 7% among the general population. With the widespread use of ultrasound (US), clinically unapparent thyroid nodule prevalence has dramatically increased with estimates at 20% to 76% in the general population. Moreover, 20% to 48% of patients with a single palpable thyroid nodule are found to have additional nodules when investigated by US.

Laser ablation therapy offer potential for the thermal destruction of soft tissue structures. The ability to deliver large doses of energy via small flexible fiberoptics makes laser therapy ideally suited for percutaneous treatment of unwanted tissue masses.

In this study we propose to treat symptomatic soft tissue thyroid masses in the head and neck region using a new FDA-cleard laser ablation system to safely and effectively debulk the tissue and therefore improve symptoms. Real time US monitoring will be performed of the ablation front to ensure complete treatment of the target lesion. All ablated regions will be followed by US with Doppler to document changes in size and vascularity. Local effects on thyroid function for thyroid mass treatment will be measured on follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented benign thyroid nodule, or cold thyroid nodule as documented by thyroid scan.
* Patient has been evaluated by endocrinology and endocrine surgery and has been deemed suitable candidate for procedure.
* The patient's nodule(s) size and number must be no larger than 5cm and a maximum of 3 nodules, respectively.
* All nodules must be greater than 1cm from the expected location of the recurrent laryngeal and vagus nerves determined under ultrasound.
* Required initial laboratory values: T3, T4. TSH, and Thyroglobulin (for treated metastatic lymph nodes)
* All patients must understand and sign a study-specific informed consent.

Exclusion Criteria:

* Thyroid mass in contact with trachea or esophagus.
* Uncontrolled coagulopathy or bleeding diathesis that cannot be corrected with FFP and platelets prior to procedure. (Platelets must be ≥ 70,000/ul.)
* Aspirin and nonsteroidal anti-inflammatory medications, antiplatelet medications, or warfarin must be discontinued prior to the procedure for a time period that is appropriate given the drug half-life and the drugs known antiplatelet activity (e.g. aspirin for 7 days and ibuprofen 24 hours). Low molecular weight heparin preparations must be discontinued 24 hours prior to procedure.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2008-02; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
The primary goal of this study is to determine the local response of laser ablation of the treated lesion and its effect on size and vascularity. The objective measures will be based on serial US with Doppler. | 12 months

SECONDARY OUTCOMES:
To assess the effects of laser ablation on thyroid function testing. An estimate of time and cost associated with LITT procedure for treatment of soft tissue thyroid nodules. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Damian Dupuy, MD, Principal Investigator — Rhode Island Hospital
Locations (1):
- Rhode Island Hospital - Department of Diagnostic Imaging Research, Providence, Rhode Island, United States